CLINICAL TRIAL: NCT06597526
Title: The Role of 18F-FDG &amp;amp;amp; 68Ga-FAPI PET/CT in the Assessment of Conversion Therapy Efficacy in Gastric Cancer with Peritoneal Metastatic
Brief Title: The Role of 18F-FDG&68Ga-FAPI PET/CT in the Assessment of Conversion Therapy Efficacy in Gastric Cancer with Peritoneal Metastasis.
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hu Jiajia, Nuclear medicine, Ruijin Hospital
Other Study IDs: RuijinH 2024-93
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Peritoneal Metastasis; Gastric Cancer
Keywords: 18F-FDG PET/CT; 68Ga-FAPI PET/CT; gastric cancer; peritoneal metastases; conversion therapy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- gastric cancer patients with peritoneal metastasis: Initial diagnosis of gastric cancer with peritoneal metastases, excluding other distant metastases

SUMMARY:
This study aims to investigate the value of 18F-FDG&68Ga-FAPI PET/CT in evaluating the outcome of conversion therapy and the prognosis of people with peritoneal metastases from gastric cancer.

DETAILED DESCRIPTION:
If the target population of the study agrees to participate in the study, we will number the participants, resume their pathology files, and collect their gender, age, phone number, height and weight information, record the participants' consultation process and the results of the tests and examinations therein. During the course of the study we will perform 18F-FDG & 68Ga-FAPI PET/CT according to the participant's stage of disease, specifically: one 18F-FDG PET/CT prior to conversion therapy and one 68Ga-FAPI PET/CT as a baseline assessment. One 18F-FDG PET/CT and one 68Ga-FAPI PET/CT were performed before the clinician assessed that the conversion therapy was ready to be completed and the conversion surgery was about to be performed, and if the participant experienced a postoperative recurrence of the disease during the study period, another 18F-FDG PET/CT and a 68Ga-FAPI PET/CT would be performed, meaning that a total of 4 PET/CTs were performed. In other words, a total of 4 PET/CT visualizations were required for all participants; 2 additional PET/CT visualizations, including 18F-FDG PET/CT and 68Ga-FAPI PET/CT, were performed if the disease recurred after the conversion surgery, and none were required for participants without recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed gastric adenocarcinoma with no history of resection of primary or metastatic lesions
2. Peritoneal metastases of gastric cancer requiring laparoscopy for definitive diagnosis without gastric outflow tract obstruction and intestinal obstruction
3. Patients voluntarily enrolled in this study by signing an informed consent form
4. Age ≥ 18 years
5. Eastern Cooperative Oncology Group (ECOG) score ≤ 2,
6. Expected life expectancy ≥ 3 months
7. Adequate organ and bone marrow function
8. Willingness to adhere to the study protocol and follow-up programme

Exclusion Criteria:

1. Signs of distant metastases other than peritoneal metastases at enrolment
2. Pregnant or breastfeeding women.
3. Patients with a history of other malignant diseases in the last 5 years, except cured skin cancer and carcinoma in situ of cervix
4. Severe mental disease, uncontrolled epilepsy, or central nervous system disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible inpatients and outpatients from Ruijin Hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-15 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Target-to-background ratio(TBR) | Baseline, preoperative assessment and time of postoperative recurrence assessment
  68Ga-FAPI and 18F-FDG uptake ratio of primary gastric lesions, peritoneal lesions and recurrent metastatic lesions to mediastinum and liver blood pool on PET/CT images.
Standardized uptake value(SUV) | Baseline, preoperative assessment and time of postoperative recurrence assessment
  SUV of 68Ga-FAPI and 18F-FDG uptake on PET/CT images for primary gastric lesions, peritoneal lesions and recurrent metastatic lesions
Evaluation the outcome of conversion therapy | Baseline and preoperative assessment
  The value of 68Ga-FAPI PET/CT and 18F-FDG PET/CT in evaluating the outcome of conversion therapy in gastric cancer with peritoneal metastasis.

SECONDARY OUTCOMES:
Progress free survival | 3 years
  Progress free survival
Overall survival | 3 years
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiao Tong University of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No